CLINICAL TRIAL: NCT00000819
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Trial to Determine the Efficacy of Prednisone Therapy in HIV-Associated Nephropathy (HIVAN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Upjohn (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 271; 11247 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; AIDS-Associated Nephropathy
Keywords: AIDS-Related Complex; Prednisone; AIDS-Associated Nephropathy
MeSH Terms: conditions — HIV Infections; AIDS-Associated Nephropathy; AIDS-Related Complex | interventions — Prednisone

INTERVENTIONS:
Drug: Prednisone

SUMMARY:
To determine the efficacy and safety of prednisone in patients with HIV-associated nephropathy. To determine the effects of prednisone on serum creatinine, urinary protein, and creatinine clearance.

HIV-associated nephropathy is characterized by heavy proteinuria, rapidly progressive renal insufficiency, and distinct nephropathologic changes. The syndrome most often occurs in patients with advanced HIV disease. Little is known about the effects of corticosteroids on the progression of HIV disease. In light of the possible beneficial effects of corticosteroids on HIV-associated nephropathy, a controlled trial using prednisone is warranted.

DETAILED DESCRIPTION:
HIV-associated nephropathy is characterized by heavy proteinuria, rapidly progressive renal insufficiency, and distinct nephropathologic changes. The syndrome most often occurs in patients with advanced HIV disease. Little is known about the effects of corticosteroids on the progression of HIV disease. In light of the possible beneficial effects of corticosteroids on HIV-associated nephropathy, a controlled trial using prednisone is warranted.

Patients are randomized to receive prednisone or placebo for 11 weeks, followed by 13 weeks of observation.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* Biopsy-confirmed glomerulosclerosis and/or mesangial proliferation within 90 days prior to study entry.
* Mild to severe renal insufficiency that is stable or worsening.
* No AIDS-defining opportunistic infections or malignancies.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Poorly controlled hypertension or diabetes mellitus.
* Peptic ulcer disease with gastrointestinal bleeding.
* Active symptomatic bacterial, protozoal, fungal, or viral infections (other than HIV disease).
* Superimposed renal disease that is due to processes other than focal glomerulosclerosis or mesangial proliferation, including but not limited to obstructive uropathy, acute tubular necrosis, and prerenal azotemia.
* Emotional problems sufficient to prevent adequate compliance with study therapy.

Concurrent Medication:

Excluded:

* IV amphotericin B.
* IV aminoglycosides.
* IV foscarnet.
* IV pentamidine.
* Trimethoprim > 200 mg/day.
* Nonsteroidal anti-inflammatory agents.
* Angiotensin converting enzyme inhibitors (benzapril, captopril, enalapril, fosinopril, lisinopril, guinapril, and ramipril) except for refractory hypertension.

Concurrent Treatment:

Excluded:

* Iodinated radiocontrast dye.

Patients with the following prior conditions are excluded:

* Active pulmonary disease on chest radiograph within 60 days prior to study entry.
* CMV retinitis on ophthalmologic evaluation within 60 days prior to study entry.
* Positive blood culture for mycobacteria 10-60 days prior to study entry.

Prior Medication:

Excluded:

* Prior corticosteroid therapy for HIVAN.
* Corticosteroid therapy for any indication within 30 days prior to study entry.
* Continuous nonsteroidal anti-inflammatory agents for more than 15 days during the 4 weeks prior to study entry.

Prior Treatment:

Excluded within 30 days prior to study entry:

* Dialysis for acute or chronic renal failure.
* Iodinated radiocontrast dye.

Required:

* Stable antiretroviral therapy with AZT alone or in combination with ddI, ddC, or d4T for at least 4 weeks unless contraindicated.
* PCP prophylaxis with TMP/SMX, pentamidine aerosol, dapsone, or atovaquone.
* MAC prophylaxis with rifabutin or clarithromycin for patients with CD4 count < 100 cells/mm3.
* Mycobacterium tuberculosis prophylaxis with isoniazid or another accepted regimen for patients with a positive or previously positive tuberculin test and for anergic patients who are known household or close contacts of infectious TB patients or who are from groups in which the prevalence of TB is 10 percent or higher.
* Investigational drugs unless exempted by protocol chair.
* Other medications unless expressly prohibited.

Active alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kalayjian R, Study Chair; Smith MC, Study Chair; Lederman M, Study Chair
Locations (8):
- United States (8):
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsf Aids Crs, San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio

REFERENCES:
- [Background] Kalayjian R, Phinney M, Austen J, Gripshover B, Carey J, Rahman M, Weigel K, Smith MC. Prednisone improves renal function in HIV-associated nephropathy (HIVAN). Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2:154